CLINICAL TRIAL: NCT00564668
Title: A 24-week, Randomised, Multi-centre, Double-blind, Parallel-group Trial to Investigate the Safety and the Efficacy of NN2000-Mix30 Compared to NN-X14Mix30 NovoRapid®30Mix) in Subjects With Type 2 Diabetes Mellitus on a Twice Daily Regimen
Brief Title: Comparison of Biphasic Insulin Aspart Produced by the NN2000 Process to Current Process to in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2000-1611
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart

SUMMARY:
This trial is conducted in Japan. The aim of this trial was to investigate the safety and efficacy of NN2000-Mix30 produced by NN2000 process compared to that of NN-X14Mix30 produced by current process in Japanese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Subjects with insulin treatment for at least 24 weeks
* Current treatment with premixed biphasic human insulin preparation for at least 12 weeks
* HbA1c lesser than or equal to 11.0%

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Proliferative retinopathy or maculopathy requiring acute treatment
* Impaired renal function
* Cardiac diseases
* Uncontrolled hypertension
* Subjects with known malignant tumour
* Total daily insulin dose greater than or equal to 100 IU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-06-19 (Actual); Primary Completion 2005-04-12 (Actual); Study Completion 2005-04-12 (Actual)

PRIMARY OUTCOMES:
Safety | During 24 weeks of treatment

SECONDARY OUTCOMES:
HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com